CLINICAL TRIAL: NCT01168635
Title: Improving Asthma Outcomes Through Spirometry Distance Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other); Boston University (Other)
Responsible Party: Principal Investigator, Rita Mangione-Smith, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13169
Record Dates: First submitted 2010-07-20; First posted 2010-07-23 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Asthma
Keywords: Asthma; Spirometry; Pediatric; Primary Health Care; Education, Distance
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Virtually-delivered spirometry quality improvement program
  Interventions: Behavioral: Spirometry 360 program - Virtually-delivered spirometry quality improvement program
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Spirometry 360 program - Virtually-delivered spirometry quality improvement program — The Spirometry 360 program includes:
  1. "Spirometry Fundamentals™: A basic guide to lung function testing," a computer-based training program that teaches primary care providers how to coach patients to produce high-quality spirometry tests and accurately interpret spirometric data;
  2. Spirometry Learning Lab: Case-based teaching of spirometry in practice guides test administrators and interpreters through clinical examples in an interactive virtual classroom setting. These sessions are led by expert clinical faculty and are archived for future reference and review;
  3. Spirometry Feedback: Tailored analysis of providers' spirometry testing sessions offers monthly individualized feedback reports by clinical experts on spirometry tests performed in the clinic.
  Arms: Intervention

SUMMARY:
Spirometry is a recommended component of asthma diagnosis and treatment in the primary care setting, yet few providers report its routine use for children with asthma. Misclassification of asthma severity occurs when assessment is based on symptoms alone. This misclassification can lead to inadequate treatment, increased morbidity, and increased healthcare utilization/cost.

The goal of this study is to test the effectiveness of a distance learning quality improvement program called Spirometry 360 developed by the interactive Medical Training Resources (iMTR) group at the University of Washington Child Health Institute. The Spirometry 360 program aims to improve care for children with asthma by enhancing provider knowledge and self-efficacy related to the use and interpretation of office-based spirometry.

DETAILED DESCRIPTION:
The Spirometry 360 program includes:

1. "Spirometry Fundamentals™: A basic guide to lung function testing," a computer-based training program that teaches primary care providers how to coach patients to produce high-quality spirometry tests and accurately interpret spirometric data;
2. Spirometry Learning Lab: Case-based teaching of spirometry in practice guides test administrators and interpreters through clinical examples in an interactive virtual classroom setting. These sessions are led by expert clinical faculty and are archived for future reference and review;
3. Spirometry Feedback: Tailored analysis of providers' spirometry testing sessions offers monthly individualized feedback reports by clinical experts on spirometry tests performed in the clinic.

This is a cluster randomized controlled trial to test the effectiveness of the Spirometry 360 program. The Spirometry 360 program will be provided to 25 primary care pediatric practices from two practice-based research networks. A separate group of 25 matched control practices recruited from these same networks will receive standard training from the equipment vendor during the study and the Spirometry 360 training program at the end of the study.

ELIGIBILITY:
Inclusion Criteria (Parent):

* Parents must have a child who has had at least one visit for asthma with a participating provider during the 12 months before the study start date
* Must have monthly access to email and the Internet
* Must have child aged 5-16 years

Inclusion Criteria (Child):

* Aged 5-16 years
* Must have access to email and the Internet

Exclusion Criteria (Parents):

* Parents with children who are outside our target age range of 5-16 years old
* Parents with children who haven't had a clinic visit for asthma care in the last year
* Parents without monthly access to the Internet

Exclusion Criteria (Child):

* Children who are outside our target age range of 5-16 years
* Children without monthly access to email and the Internet

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 660 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Healthcare utilization | Assessed monthly for 1 year
  Parent report of number of Emergency Room/Emergency Department (ER/ED) visits, unplanned outpatient visits, and number of hospitalizations due to asthma in the last month.
Cost of asthma care | Every 6 months
  Cost in inflation-adjusted dollars for unplanned healthcare utilization due to asthma exacerbation, including unplanned office visits, ED visits, and asthma-related hospitalization.
Asthma-specific health-related quality of life | Every 6 months
  Parent report of child's asthma-specific health-related quality of life. Measured using )Pediatric Quality of Life Inventory (PedsQL)(TM) 3.0 Short Form (SF)-22 Asthma Module. The tool consists of an 11-item symptoms scale and an 11-item treatment problems scale.

SECONDARY OUTCOMES:
Acceptable spirometry testing sessions | Assessed monthly for 1 year
  Monthly proportion of spirometry tests performed by enrolled practices with acceptable quality grades during intervention.
Appropriate prescription of controller therapy | Assessed monthly for 1 year
  Parent/child report asthma symptoms and unplanned health care utilization consistent with persistent/uncontrolled asthma AND patient has been prescribed a controller medication.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mangione-Smith, MD, MPH, Principal Investigator — Seattle Children's Hospital/University of Washington
Locations (4):
- United States (4):
  - Slone Center Office-based Research Network (SCOR) - Boston University, Boston, Massachusetts
  - Seattle Children's Hospital Research Institute, Seattle, Washington
  - Child Health Institute - Unversity of Washington, Seattle, Washington
  - Puget Sound Pediatric Research Network, Seattle, Washington

REFERENCES:
- See also: Site for primary care physicians to learn about Spirometry — http://www.spirometrytraining.org/